CLINICAL TRIAL: NCT06960330
Title: Wearable Biofeedback Devices for Remote Physiotherapy and Rehabilitation for Elderly Patients Suffering From Arthritis and Fibromyalgia
Brief Title: Wearable Biofeedback Devices for Remote Physiotherapy and Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Advanced Education & Research Center (Other)
Responsible Party: Principal Investigator, Shamoon Noushad, Professor, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WBD-RPRAEF-2025
Record Dates: First submitted 2025-04-19; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Arthritis; Fibromyalgia; Chronic Pain
MeSH Terms: conditions — Arthritis; Fibromyalgia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups:
  Intervention Group - receives wearable biofeedback devices with guided exercises and virtual physiotherapy.
  Control Group - receives standard physiotherapy exercises without biofeedback.
Masking Description: Due to the nature of the intervention (wearable devices and virtual consultations), blinding of participants and care providers is not feasible. This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will receive wearable biofeedback devices integrated with guided exercise routines and virtual physiotherapy consultations over a set period (e.g., 12 weeks). The devices will provide real-time physiological monitoring and feedback, including heart rate variability (HRV), to guide home-based rehabilitation.
  Intervention Name:
  Wearable Biofeedback + Virtual Physiotherapy
  Intervention Type:
  Device (or Behavioral, depending on how the registry classifies it)
  Intervention Description:
  Participants will use wearable devices designed to monitor physiological parameters and provide real-time feedback during exercises. The intervention includes remote guidance from physiotherapists via virtual consultations.
  Interventions: Other: Wearable Biofeedback + Virtual Physiotherapy
- Control Group (Active Comparator): Participants in this group will perform a standard physiotherapy exercise regimen without any wearable biofeedback device or virtual consultation support.
  Intervention Name:
  Standard Physiotherapy Exercises
  Intervention Type:
  Behavioral
  Intervention Description:
  Participants will be given printed or video instructions for standard physiotherapy exercises commonly used for arthritis and fibromyalgia management, without any digital monitoring or remote guidance.
  Interventions: Other: Standard Physiotherapy Exercises

INTERVENTIONS:
Other: Wearable Biofeedback + Virtual Physiotherapy — Participants will use wearable devices designed to monitor physiological parameters and provide real-time feedback during exercises. The intervention includes remote guidance from physiotherapists via virtual consultations.
  Arms: Intervention Group
Other: Standard Physiotherapy Exercises — Participants will be given printed or video instructions for standard physiotherapy exercises commonly used for arthritis and fibromyalgia management, without any digital monitoring or remote guidance.
  Arms: Control Group

SUMMARY:
This study evaluates the effectiveness of wearable biofeedback devices in improving pain, mobility, and rehabilitation outcomes in elderly patients with arthritis and fibromyalgia in Karachi, Pakistan. In a randomized controlled trial involving 120 participants, one group will use biofeedback-integrated devices with guided exercises and virtual consultations, while the control group receives standard physiotherapy. The results will inform the potential of digital health solutions to improve accessibility and outcomes in remote rehabilitation for chronic pain management.

DETAILED DESCRIPTION:
Arthritis and fibromyalgia are common chronic musculoskeletal conditions among the elderly population, contributing to significant pain, reduced mobility, and diminished quality of life. In urban centers like Karachi, Pakistan, access to consistent and effective physiotherapy is often hindered by mobility limitations and inadequate healthcare infrastructure. This randomized controlled trial (RCT) investigates the efficacy of wearable biofeedback devices as an innovative approach to address these challenges.

A total of 120 elderly participants diagnosed with arthritis and/or fibromyalgia will be enrolled and randomized into two groups (60 participants per group). The intervention group will receive wearable biofeedback devices that monitor physiological parameters such as heart rate variability (HRV) and provide real-time feedback during guided home-based exercises, complemented by virtual physiotherapy consultations. The control group will follow standard physiotherapy exercise routines without biofeedback or virtual support.

Primary outcome measures include pain intensity (measured using a standardized pain scale), functional mobility (assessed via timed mobility tests), and joint range of motion. Secondary outcomes will assess heart rate variability, patient adherence to exercise protocols, and changes in psychological well-being.

This study seeks to determine whether wearable biofeedback can enhance rehabilitation outcomes, promote exercise adherence, and offer a viable, accessible alternative to conventional physiotherapy. If successful, the intervention could transform chronic pain management and rehabilitation strategies for aging populations, especially in resource-constrained urban environments.

ELIGIBILITY:
Inclusion Criteria:

Elderly adults aged 60-80 years diagnosed with arthritis or fibromyalgia.

Experiencing moderate to severe pain and mobility limitations.

No recent surgical interventions or contraindications for physiotherapy.

Access to smartphones and internet connectivity for remote monitoring.

Exclusion Criteria:

Patients with severe cognitive impairments affecting adherence to rehabilitation.

Presence of comorbidities that contraindicate physiotherapy (e.g., severe cardiac conditions).

Lack of access to digital devices required for remote monitoring.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-06 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (VAS Score) | Baseline, Week 6, Week 12
  Pain intensity will be measured using the Visual Analog Scale (VAS), a 10-cm horizontal line where participants mark their perceived pain level from 0 (no pain) to 10 (worst imaginable pain).
Functional Mobility (Timed Up and Go Test) | Baseline, Week 6, Week 12
  Functional mobility will be assessed using the Timed Up and Go (TUG) Test. Participants will be timed as they rise from a chair, walk 3 meters, turn, return, and sit down again.
Range of Motion (Goniometry) | Baseline, Week 6, Week 12
  Joint range of motion will be measured using a goniometer to assess changes in movement capacity of affected joints (e.g., knees, shoulders).

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | Baseline, Week 6, Week 12
  HRV will be evaluated using time-domain (e.g., RMSSD) and frequency-domain (e.g., LF/HF ratio) metrics recorded by wearable devices.
Patient Adherence | Throughout the 12-week intervention
  Adherence to prescribed exercises will be monitored through device usage logs, measuring frequency and duration of engagement with the intervention.
Change in Depression Severity (Beck Depression Inventory Score) | Baseline, Week 12
  The BDI score ranges from 0 to 63. Higher scores indicate more severe depressive symptoms.
System Usability and Patient Satisfaction | Week 12
  The SUS consists of 10 items, each rated on a 5-point Likert scale (from Strongly Agree to Strongly Disagree). The total score ranges from 0 to 100. A higher score indicates better usability and user satisfaction.
Change in Quality of Life (SF-36 Health Survey Score) | Baseline, Week 12
  The SF-36 consists of 8 scaled scores (0-100). Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Basit Ansari, Ph.D., Study Director — University of Karachi
Locations (1):
- University of Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akhter E, Bilal S, Kiani A, Haque U. Prevalence of arthritis in India and Pakistan: a review. Rheumatol Int. 2011 Jul;31(7):849-55. doi: 10.1007/s00296-011-1820-3. Epub 2011 Feb 18. PMID 21331574
- [Result] Dagnino APA, Campos MM. Chronic Pain in the Elderly: Mechanisms and Perspectives. Front Hum Neurosci. 2022 Mar 3;16:736688. doi: 10.3389/fnhum.2022.736688. eCollection 2022. PMID 35308613
- [Result] Danilin LK, Spindler M, Soros P, Bantel C. Heart rate and heart rate variability in patients with chronic inflammatory joint disease: the role of pain duration and the insular cortex. BMC Musculoskelet Disord. 2022 Jan 21;23(1):75. doi: 10.1186/s12891-022-05009-1. PMID 35062938
- [Result] Dudarev V, Barral O, Radaeva M, Davis G, Enns JT. Night time heart rate predicts next-day pain in fibromyalgia and primary back pain. Pain Rep. 2024 Feb 1;9(2):e1119. doi: 10.1097/PR9.0000000000001119. eCollection 2024 Apr. PMID 38322354